CLINICAL TRIAL: NCT00798304
Title: An Open Label, Randomized, Phase 1/2 Trial Of The Safety, Tolerability, And Immunogenicity Of Meningococcal Group B Rlp2086 Vaccine In Healthy Infants
Brief Title: Study Evaluating Safety, Tolerability, and Immunogenicity of Meningococcal B Vaccine in Healthy Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following program review within Pfizer, decision was made not to go ahead with this study. This study is cancelled
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6108K2-2000; B1971008 (Other: Alias Study Number); 2008-001457-18 (EudraCT Number)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningococcal B vaccine; infants; safety; immunogenicity
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Dose level 1 of meningococcal B rLP2086 vaccine and routine childhood vaccines
  Interventions: Biological: meningococcal B rLP2086 vaccine; Biological: Routine age appropriate childhood vaccines
- 2 (Experimental): Dose level 2 of meningococcal B rLP2086 vaccine and routine childhood vaccines
  Interventions: Biological: meningococcal B rLP2086 vaccine; Biological: Routine age appropriate childhood vaccines
- 3 (Experimental): Control group
  Interventions: Biological: Routine age appropriate childhood vaccines

INTERVENTIONS:
Biological: meningococcal B rLP2086 vaccine — vaccination
  Arms: 1
Biological: Routine age appropriate childhood vaccines — vaccination
  Arms: 1
Biological: meningococcal B rLP2086 vaccine — vaccination
  Arms: 2
Biological: Routine age appropriate childhood vaccines — vaccination
  Arms: 2
Biological: Routine age appropriate childhood vaccines — vaccination
  Arms: 3

SUMMARY:
The primary purpose of this study is to evaluate the safety and immunogenicity of an investigational meningococcal B vaccine in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Investigators should always use good clinical judgment in considering a subject's overall fitness for trial participation. In addition, any condition that in the opinion of the investigator may interfere with the evaluation of study objectives should be carefully considered prior to enrolling subjects.
* Male or female subjects aged 2 months (42 to 98 days of age) at the time of enrollment.
* Available for the entire consented period and whose parent/legal guardian can be reached by telephone.
* Healthy infant as determined by medical history, physical examination, and judgment of the investigator.
* Parent/legal guardian must be able to complete all relevant study procedures during study participation.

Exclusion Criteria:

* Previous vaccination with licensed or investigational vaccines: meningococcal B, meningococcal C, pneumococcal, Hib, diphtheria, tetanus, acellular pertussis, poliovirus, rotavirus, varicella, measles, mumps, or rubella.

Any of the following illnesses/conditions that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study:

* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with meningococcal B, meningococcal C, pneumococcal, Hib, diphtheria, tetanus, acellular pertussis, Hepatitis B (HBV), poliovirus, rotavirus, varicella, measles, mumps, or rubella.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* Known or suspected immune deficiency or suppression.
* History of culture-proven invasive disease caused by N meningitidis or Neisseria gonorrhoea.
* Major known congenital malformation or serious chronic disorder.
* Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorder such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorder.

Does not include resolving syndromes due to birth trauma such as Erb palsy.

* Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies).
* Received any investigational drugs, vaccines or devices (aside from those specified in the protocol) within 4 weeks before administration of the first dose of test article or at any time throughout the study.
* Participation in purely observational studies is acceptable.
* Infant who is a direct descendant (child, grandchild) of the study site personnel.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Spain (7):
  - Clínica Mediterráneo, Almería, Almeria
  - Hospital Clinico Universitario de Santiago, Santiado de Compostela, La Coruña
  - Hospital Gral. Gregorio Maranon, Madrid, Madrid
  - Hospital 12 de Octubre Materno-Infantil Unidad de Lactantes, Madrid, Madrid
  - Hospital Universitario de Mostóles, Mostóles, Madrid
  - Hospital Virgen del Camino, Pamplona, Navarre
  - Hospital Xeral de Vigo, Vigo

REFERENCES:
- [Derived] Martinon-Torres F, Gimenez-Sanchez F, Bernaola-Iturbe E, Diez-Domingo J, Jiang Q, Perez JL. A randomized, phase 1/2 trial of the safety, tolerability, and immunogenicity of bivalent rLP2086 meningococcal B vaccine in healthy infants. Vaccine. 2014 Sep 8;32(40):5206-11. doi: 10.1016/j.vaccine.2014.07.049. Epub 2014 Jul 29. PMID 25077420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, participants were to receive recombinant lipoprotein 2086 (rLP2086) vaccine at 2, 4, 6 and 12 months of age. Due to premature termination of study, only single dose of 20 or 60 microgram (mcg) of rLP2086 vaccine was administered at 2 months and planned treatments of rLP2086 vaccine 120 mcg and 200 mcg were not administered.
Groups:
- Control: Routine childhood vaccines (InfanrixHexa, Meningitec, Prevenar and Rotarix) according to local practice.
- rLP2086 20 mcg: Recombinant lipoprotein 2086 (rLP2086) 20 microgram (mcg) vaccine along with routine childhood vaccines according to local practice.
- rLP2086 60 mcg: rLP2086 60 mcg vaccine along with routine childhood vaccines according to local practice.
Period: Overall Study
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Started | 14 | 22 | 10
Completed | 0 | 0 | 0
Not Completed | 14 | 22 | 10
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Discontinuation by Sponsor | 14 | 21 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg | Total
Number analyzed (Participants) | 14 | 22 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: days] | 63.6 (11.57) | 64.0 (10.02) | 71.6 (11.35) | 65.5 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 4 | 22
  Male | 8 | 10 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least 1:4 rLP2086-specific Serum Bactericidal Assay (SBA) Titer to 1 Subfamily A Strain and 1 Subfamily B Strain
Time Frame: 1 month after Dose 3
Population: Results were not reported for this outcome measure because the study was terminated prior to the first scheduled post-vaccination blood draw and no immunogenicity data were collected.
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Serum Bactericidal Assay (SBA) Geometric Mean Titers (GMTs) for 1 Subfamily A Strain and 1 Subfamily B Strain
Time Frame: 1 month after Dose 2, Dose 3; before Dose 4
Population: as for outcome 1
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving at Least 1:4, 1:8, 1:16, 1:32, 1:64, 1:128 rLP2086-specific SBA Titer to 1 Subfamily A Strain and 1 Subfamily B Strain
Time Frame: 1 month after Dose 2, Dose 3; before Dose 4
Population: as for outcome 1
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Percentage of Participants Achieving Response >=1:4 for Additional Meningococcal Serogroup B (MnB) Test Strain-specific SBA Titer
Time Frame: 1 month after Dose 2, Dose 3; before Dose 4; 1, 6, 12, 18, 24, 36, 48 months after Dose 4
Population: as for outcome 1
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Percentage of Participants Achieving SBA Titer Levels >=1:4, >=1:8, >=1:16, >=1:32, >=1:64 and >=1:128 for Additional MnB Test Strains
Time Frame: 1 month after Dose 2, Dose 3; before Dose 4; 1, 6, 12, 18, 24, 36, 48 months after Dose 4
Population: as for outcome 1
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Serum Bactericidal Assay (SBA) GMTs for Additional MnB Test Strains
Time Frame: 1 month after Dose 2, Dose 3; before Dose 4; 1, 6, 12, 18, 24, 36, 48 months after Dose 4
Population: as for outcome 1
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: From signing of informed consent form to completion of study (up to 2 years)
Measure: Number; unit: percentage of participants
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Number analyzed (Participants) | 14 | 22 | 10
percentage of participants | 21.4 | 31.8 | 20.0

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study (up to 2 years)
Arm/Group | Control | rLP2086 20 mcg | rLP2086 60 mcg
Serious Adverse Events (participants affected / at risk) | 0/14 | 4/22 | 1/10
Other Adverse Events (participants affected / at risk) | 3/14 | 4/22 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=14) | rLP2086 20 mcg (N=22) | rLP2086 60 mcg (N=10)
Bronchitis (Infections and infestations) | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=14) | rLP2086 20 mcg (N=22) | rLP2086 60 mcg (N=10)
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Immunogenicity results were not reported because the study was terminated due to the reactogenicity profile of the vaccine in infants prior to the first scheduled post-vaccination blood draw and no immunogenicity data were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.